CLINICAL TRIAL: NCT01074931
Title: Clinical, Virological and Safety Outcomes of a Lopinavir/Ritonavir-Based Regimen in HIV-1 Infected Patients in Routine Clinical Use in China: A Multicenter Post-Marketing Observational Study
Brief Title: Clinical, Virological and Safety Outcomes of a Lopinavir/Ritonavir-Based Regimen in HIV-1 Infected Patients in Routine Clinical Use in China
Status: Completed | Type: Observational
Sponsor: Abbott (Industry)
Responsible Party: Yue Kang, Abbott China
Other Study IDs: P10-398
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2011-08-03 (Estimated); Last update posted 2011-08-03 (Estimated); Status verified 2011-07

CONDITIONS: HIV-1 Infections
Keywords: Lopinavir/ritonavir
MeSH Terms: interventions — Lopinavir; Ritonavir; lopinavir-ritonavir drug combination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Lopinavir/ritonavir group: This study is a non-interventional, observational study in which lopinavir/ritonavir is prescribed in the usual manner in accordance with the terms of China market authorization with regards to dose, population and indication. It is planned to enroll approximately 100 patients in total.
  Interventions: Drug: Lopinavir/ritonavir (Kaletra)

INTERVENTIONS:
Drug: Lopinavir/ritonavir (Kaletra) — Lopinavir/ritonavir(LPV/r) is an HIV protease inhibitor (PI) that is co-formulated with lopinavir and ritonavir. Lopinavir is an inhibitor of the HIV-1 and HIV-2 proteases. As co-formulated in LPV/r, ritonavir inhibits the CYP3A-mediated metabolism of lopinavir, thereby providing increased plasma levels of lopinavir.
  The assignment of the patient to a lopinavir/ritonavir - containing regimen is not decided in advance by this protocol but falls within current practice and the prescription of lopinavir/ritonavir is clearly separated from the decision to include the patient in this study.
  Other Names: lopinavir/ritonavir; Kaletra

SUMMARY:
This post-marketing observational study is conducted for obtaining data on clinical, biological and virological outcomes, compliance and tolerability of using a lopinavir/ritonavir (LPV/r) -containing regimen for the treatment of naïve or experienced patients infected with human immunodeficiency virus type 1 (HIV-1) in China.

Although LPV/r is frequently used world-wide, the evaluation of the outcomes, compliance, and tolerance of anti-HIV strategies in real life is still a major challenge in the management of HIV-infected patients who are on a life-long therapy, especially in China.

This study will help to develop effectiveness and safety profile of the lopinavir/ritonavir containing regimen in Chinese HIV-1 infected patients, provide more choices of anti-HIV-1 strategies to Chinese experts and benefits Chinese HIV-1 infected patients.

DETAILED DESCRIPTION:
It is planned to enroll approximately 100 patients in total. This will be a multicenter post-marketing observational study in China mainland.

Each patient will be observed during his/her lopinavir/ritonavir - containing treatment regimen for a maximum period of 18 months.

If the physician decides to permanently discontinue lopinavir/ritonavir before the end of the planned observational period of 18 months, the reason for the discontinuation and the new treatment regimen prescribed will be documented. The next routine follow-up visit will be the termination visit for this patient in this study.

This post-marketing observational study will be conducted in a prospective, single-arm, multicenter format.

As this study is observational in nature, its follow-up is not interventional and is left to the judgment of each physician within the 18-month period, which defines the survey for each patient. For indicative purpose, follow-up of patients should enable approximately 4 patient visits during this period. These visits will take place at average intervals of 6 months, apart from the first visit following inclusion (usually at the end of the first 3 treatment months) and apart from visits required because of an intercurrent event. If treatment with lopinavir/ritonavir is discontinued, standard practice is to review the patient after a period of 3 months.

For these reasons, the most likely visits are defined as "V1", "V2", "V3", "V4" although numbers and dates will depend only on the decision of the physician. As a result, failure to meet these suggested dates will not constitute a deviation of the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Patients infected by HIV-1 who are over 18 years old
* Patients who belong to one of the following cohorts:

  * Antiretroviral naïve patients
  * Antiretroviral experienced patients, irrespective to their immune and viral status and current antiretroviral therapy

Exclusion Criteria:

* Patients who have been treated with lopinavir/ritonavir
* Patients who are being treated or will be treated with drugs at risk of interactions with lopinavir/ritonavir
* Patients who are not tolerant to lopinavir/ritonavir
* Patients who have uncontrolled AIDS defining disease
* Patients participating in another clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2008-04; Primary Completion 2010-05 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian LI, MD, Study Chair — Abbott (China)
Locations (5):
- China (5):
  - Site Reference ID/Investigator# 7244, Guangdong
  - Site Reference ID/Investigator# 27865, Kunming
  - Site Reference ID/Investigator# 27864, Shanghai
  - Site Reference ID/Investigator# 27863, Shenzhen
  - Site Reference ID/Investigator# 27866, Zhengzhou

RESULTS

PARTICIPANT FLOW:
Groups:
- Lopinavir/Ritonavir Group: Adult participants with HIV-1 infection taking lopinavir/ritonavir
Period: Overall Study
Arm/Group | Lopinavir/Ritonavir Group
Started | 98
Completed | 92
Not Completed | 6
Not completed — Economic reasons | 1
Not completed — Death | 5

BASELINE CHARACTERISTICS:
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 98
Age Continuous [Mean (Standard Deviation); unit: years] | 39.86 (10.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 71
Region of Enrollment [Number; unit: participants]
  China | 98
Age at HIV-1 Diagnosis [Mean (Standard Deviation); unit: years] — The mean age at which participants were diagnosed with HIV-1, based on 97 participants.
  years | 36.35 (10.89)
Participant Classification [Number; unit: Participants] — Participants were classified as either treatment-naive or treatment experienced.
  Participants
    Treatment-experienced | 90
    Treatment-naive | 8
WHO Clinical Staging [Number; unit: Participants] — Participants were staged according to the World Health Organization (WHO) clinical classification of established HIV infection: Stage 1 (asymptomatic), Stage 2 (mild symptoms), Stage 3 (advanced symptoms), and Stage 4 (severe symptoms).
  Participants
    Stage 1 (asymptomatic) | 8
    Stage 2 (mild symptoms) | 22
    Stage 3 (advanced symptoms) | 32
    Stage 4 (severe symptoms) | 36
Body Weight [Mean (Standard Deviation); unit: kilograms] — Participant body weight at study entry.
  kilograms | 56.91 (11.14)
Lipodystrophy [Number; unit: Participants] — The presence and severity of lipodystrophy (abnormal body fat distribution) at study entry.
  Participants
    Lipodystrophy not present | 56
    Mild lipodystrophy present | 30
    Moderate lipodystrophy present | 11
    Severe lipodystrophy present | 1
Antiretroviral Treatment within Previous 6 Months [Number; unit: Particpants] — Whether or not the participant had antiretroviral treatment within 6 months prior to study entry.
  Particpants
    Yes | 89
    No | 8
    Not reported | 1
Other Chronic Diseases Present [Number; unit: participants] — Whether or not the participant had a chronic disease that had developed previously or was identified at study entry.
  participants
    No | 67
    Yes | 29
    Not reported | 2

OUTCOME MEASURES:

1. Primary Outcome: Evolution of the HIV Viral Response
Description: The protocol recommended that HIV viral load tests be performed at baseline and each study visit. Test results indicate the number of HIV-1 ribonucleic acid (RNA) copies per milliliter (mL). The number of participants who underwent testing and had detectable levels (greater than 50 copies/mL) or undetectable levels (less than 50 copies/mL) are presented by subgroup. Study visits were to occur at approximately 3, 6, 12, and 18 months after starting treatment. The exact dates of each visit depended on the physician's judgment, so data are reported for Visits 1 through 4 rather than by month.
Time Frame: Month 3, 6, 12, 18
Population: All participants who took at least one dose of lopinavir/ritonavir and had HIV viral load testing.
Measure: Number; unit: participant
Groups:
- Lopinavir/Ritonavir: Treatment-naive: The subgroup of participants who had not received prior antiretroviral drug therapy.
- Lopinavir/Ritonavir: Treatment-experienced: The subgroup of participants who had previously received antiretroviral drug therapy.
Arm/Group | Lopinavir/Ritonavir: Treatment-naive | Lopinavir/Ritonavir: Treatment-experienced
Number analyzed (Participants) | 1 | 66
participant
  Viral load detectable at Baseline | 0 | 51
  Viral load detectable at Visit 1 | 0 | 3
  Viral load detectable at Visit 2 | 0 | 12
  Viral load detectable at Visit 3 | 0 | 5
  Viral load detectable at Visit 4 | 0 | 5
  Viral load undetectable at Baseline | 1 | 15
  Viral load undetectable at Visit 1 | 0 | 22
  Viral load undetectable at Visit 2 | 0 | 39
  Viral load undetectable at Visit 3 | 1 | 47
  Viral load undetectable at Visit 4 | 0 | 25

2. Primary Outcome: Evolution of CD4 Count
Description: The evolution of participants' CD4-positive (CD4+) T-lymphocyte counts after starting the lopinavir/ritonavir-containing regimen was to be assessed by measuring the number of CD4+ cells at baseline and each subsequent study visit. CD4+ count results are reported as the number of CD4+ cells per cubic millimeter (cmm). Study visits were to occur at approximately 3, 6, 12, and 18 months after starting treatment. The exact dates of each visit depended on the physician's judgment, so data are reported for Visits 1 through 4 rather than by month.
Time Frame: Month 3, 6, 12, 18
Population: Includes all participants taking at least one dose of lopinavir/ritonavir who had CD4+ count results at each particular time point.
Measure: Mean (Standard Deviation); unit: cells per cmm
Arm/Group | Lopinavir/Ritonavir: Treatment-naive | Lopinavir/Ritonavir: Treatment-experienced
Number analyzed (Participants) | 8 | 90
cells per cmm
  CD4+ count at Baseline | 101.00 (107.94) | 249.03 (196.40)
  CD4+ count at Visit 1 | 136.67 (85.20) | 285.96 (164.05)
  CD4+ count at Visit 2 | 200.57 (123.25) | 317.10 (180.26)
  CD4+ count at Visit 3 | 200.00 (112.56) | 378.56 (198.35)
  CD4+ count at Visit 4 | 239.00 (124.40) | 413.77 (209.96)

3. Primary Outcome: Evolution of the Tolerance Issues
Description: At each study visit, treating physicians evaluated participants and used their clinical judgment to determine if they were tolerating the lopinavir/ritonavir-containing regimen. Study visits were to occur at approximately 3, 6, 12, and 18 months after starting treatment. The exact dates of each visit depended on the physician's judgment, so data are reported for Visits 1 through 4 rather than by month.
Time Frame: Month 3, 6, 12, 18
Population: All participants taking at least one dose of lopinavir/ritonavir.
Measure: Number; unit: Participants
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 98
Participants
  Lopinavir/ritonavir not tolerated at Visit 1 | 2
  Lopinavir/ritonavir not tolerated at Visit 2 | 0
  Lopinavir/ritonavir not tolerated at Visit 3 | 0
  Lopinavir/ritonavir not tolerated at Visit 4 | 0

4. Secondary Outcome: Number of Participants Who Missed Doses, Interrupt or Discontinue Regimen, and Experience Changes in Dosage or of Combination Regimen
Description: Visits were to occur at approximately 3, 6, 12, and 18 months after starting treatment. The frequency with which each participant forgot to take their medication since the last visit and discontinuations of treatment and the reasons were documented at each visit and are summarized. The number of participants changing from lopinavir/ritonavir soft gel capsule to tablet are also presented. The exact dates of each visit depended on the physician's judgment, so data are reported for Visits 1 through 4 rather than by month. Note: participants may have had multiple missed doses or therapy changes.
Time Frame: Month 3, 6, 12, 18
Population: All participants who took at least one dose of lopinavir/ritonavir.
Measure: Number; unit: Participants
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 98
Participants
  Total Missed Doses | 49
  a) Missed doses reported at Visit 1 | 9
  b) Missed doses reported at Visit 2 | 13
  c) Missed doses reported at Visit 3 | 17
  d) Missed doses reported at Visit 4 | 10
  Discontinued lopinavir/ritonavir therapy | 6
  a) Discontinued due to serious adverse event | 5
  b) Discontinued due to economic reasons | 1
  Interrupted lopinavir/ritonavir therapy | 4
  a) Interrupted due to adverse event | 2
  b) Required treatment with prohibited medication | 1
  c) Away because of work | 1
  Therapy change: Switch from capsule to tablet | 51
  a) Switch from capsule to tablet at Visit 1 | 35
  b) Switch from capsule to tablet at Visit 2 | 12
  c) Switch from capsule to tablet at Visit 3 | 4
  d) Switch from capsule to tablet at Visit 4 | 0

5. Secondary Outcome: Adverse Events Observed and Development of Lipodystrophy Lesion and Their Locations
Description: The types of adverse events reported are summarized. The presence of lipodystrophy (abnormal body fat distribution) and its location was to be recorded. However, due to an oversight, there was not a place to record the location of lipodystrophy on the case report form. Doctors used clinical judgment to rate lipodystrophy in treatment-experienced participants. Study visits were to occur at approximately 3, 6, 12, and 18 months after starting treatment. The exact dates of each visit depended on the physician's judgment, so data are reported for Visits 1 through 4 rather than by month.
Time Frame: Month 3, 6, 12, 18
Population: The adverse event population includes all participants who took at least one dose of lopinavir/ritonavir (98). Lipodystrophy evaluations were performed in treatment-experienced participants (90), not treatment-naive participants (8).
Measure: Number; unit: Participants
Arm/Group | Lopinavir/Ritonavir Group
Number analyzed (Participants) | 98
Participants
  Non-serious adverse events | 1
  Serious adverse events | 8
  Lipodystrophy: Visit 1 evaluation | 90
  a) Improved | 24
  b) Unchanged | 65
  c) Worsened | 1
  Lipodystrophy: Visit 2 evaluation | 88
  a) Improved | 8
  b) Unchanged | 78
  c) Worsened | 2
  Lipodystrophy: Visit 3 evaluation | 87
  a) Improved | 8
  b) Unchanged | 79
  c) Worsened | 0
  Lipodystrophy: Visit 4 evaluation | 84
  a) Improved | 9
  b) Unchanged | 75
  c) Worsened | 0

6. Secondary Outcome: The Duration on Treatment Until Development of an Adverse Event Leading to Treatment Discontinuation or Until Escape From Treatment
Description: As so few participants withdrew from lopinavir/ritonavir treatment, durations of lopinavir/ritonavir therapy required for 25 percent, 50 percent and 75 percent of participants could not be established. The numbers of participants in each subgroup who discontinued from treatment due to an adverse event are presented.
Time Frame: Month 3, 6, 12, 18
Population: All participants who took at least one dose of lopinavir/ritonavir.
Measure: Number; unit: Participants
Groups:
- Lopinavir/Ritonavir Group: Treatment-naive: The subgroup of participants who had not received prior antiretroviral drug therapy.
- Lopinavir/Ritonavir Group: Treatment-experienced: The subgroup of participants who had previously received antiretroviral drug therapy.
Arm/Group | Lopinavir/Ritonavir Group: Treatment-naive | Lopinavir/Ritonavir Group: Treatment-experienced
Number analyzed (Participants) | 8 | 90
Participants | 1 | 5

ADVERSE EVENTS:
Time Frame: All adverse events that occurred during the course of the study were reported in detail on case report forms. Adverse events occurring during the study were reported up to 30 days or 5 half-lives after the last dose of lopinavir/ritonavir.
Description: The safety population included all participants who took at least 1 dose of lopinavir/ritonavir.
Arm/Group | Lopinavir/Ritonavir Group
Serious Adverse Events (participants affected / at risk) | 8/98
Other Adverse Events (participants affected / at risk) | 1/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lopinavir/Ritonavir Group (N=98)
Hypoproteinemia (Metabolism and nutrition disorders) | 1 (1)
Liver and kidney syndromes (Hepatobiliary disorders) | 1 (1)
Hepatocirrhosis (Hepatobiliary disorders) | 1 (1)
Serious hepatitis (Hepatobiliary disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chest distress (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Severe pneumonia (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Bone fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Port colored urine (Renal and urinary disorders) | 1 (1)
Infections (Immune system disorders) | 2 (2)
Tuberculosis (Immune system disorders) | 2 (2)
Fever (General disorders) | 2 (2)
Death (General disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Wasting syndrome (General disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Hepatic encephalopathy (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lopinavir/Ritonavir Group (N=98)
Hyperlipidemia (Metabolism and nutrition disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The location of lipodystrophy was not summarized as there was not a place to record the information on the case report form. Too few participants withdrew from treatment to conduct planned analyses of duration to adverse event(s)/discontinuation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Abbott requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. Abbott requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if Abbott needs to secure patent or proprietary protection.